CLINICAL TRIAL: NCT03864289
Title: Parent Skills Training for Families of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDEK-PST-2019
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent skills training (Experimental): Parents of children with autism spectrum disorder attend the parental training course once a week, and there was a total of eight courses with each course lasting 3 hours.
  Interventions: Behavioral: Parent skills training

INTERVENTIONS:
Behavioral: Parent skills training — Parents of children with autism spectrum disorder attend the parental training course once a week, and there was a total of eight courses with each course lasting 3 hours
  Other Names: PST

SUMMARY:
The study is focused on helping parents master the basic intervention skills and evaluate the effectiveness of this parental training style for children with autism spectrum disorder in China.

DETAILED DESCRIPTION:
The investigators designed a set of parental training curriculum about early intervention.

The curriculum consists of three units: (1) Delivery of theoretical intervention knowledge and analysis of successful training cases; (2) Commenting and making suggestion on parent-child interaction videos; (3) Demonstration of intervention skills and practice .The contents of the curriculum involved setting up an environment, developing objectives (verbal communication, non-verbal communication, social interaction, imitation, fine motor skills, etc.), designing activities, dealing with challenging behavior. This study will help parents master the basic intervention skills(how to set up an environment, develop objectives, design activities, deal with challenging behavior, etc) . At last the investigators will evaluate the effectiveness of this parental training style for children with autism spectrum disorder in China.

ELIGIBILITY:
Inclusion Criteria:

* Children with ASD or high risk for autism;
* Han ethic;
* Parents were at least middle school educated, and agreed to do at least 20 hours per week of planned practice activities with the child in daily life.

Exclusion Criteria:

* Children with Syndromic ASD caused by known genetic defects or inherited metabolic diseases , such as Rett Syndrome, Fragile X Syndrome, Angelman Syndrome, Prader-Willi Syndrome, tuberous sclerosis;
* Visual, auditory and physical disabilities;
* Complication with other serious chronic diseases, such as liver and kidney failure, connective tissue diseases, tumors.

Ages: 18 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline average score of the Interaction Fidelity Rating System at 8 weeks | From enrollment to end of training（8 week）. The score will be measured at the following time point: enrollment,end of training.
  The Interaction Fidelity Rating System is used to evaluate the quality of the parent mastery of intervention skills and the quality of interaction. It's a 5-point rating system (1-5) of 11 items. Parent fidelity is rated from the parent-child interaction videos by trainers. The investigators take the average score of the 11 items as a result. The highest score is 5 and the lowest is 1. The higher the score is, the better intervention skills the parents had.
  The 5-point rating system:
  1 - the strategy is not demonstrated or inappropriately applied.
  2- the strategy is used somewhat appropriately at times.
  3 - appropriate and accurate implementation of the strategy occurs up to 50% of the time.
  4 - appropriate and accurate implementation of the strategy occurs up to 80% of the time.
  5- Strategies are applied appropriately in 80-100% of opportunities.
Change from baseline correct answer rate of the Questionnaire on Awareness and Knowledge of Interventions about Autism at 8 weeks | From enrollment to end of training（8 week）. The correct rate will be measured at the following time point: enrollment, end of training.
  The Questionnaire on Awareness and Knowledge of Interventions about Autism includes 11 questions. Parents filled in the questionnaire. The investigators take the correct rate as a result. If all the 11 questions were answered correctly, the correct rate would be 100%. The highest correct rate is 100% and the lowest is 0%.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Xu, Doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China